CLINICAL TRIAL: NCT06789653
Title: Investigating Cellular Senescence and Organ Aging in Breast Cancer Patients Undergoing Adjuvant Chemotherapy: A Novel Approach Utilizing Organ Specific Age Proteomics
Brief Title: A Novel Approach Utilizing Organ Specific Age Proteomics
Status: Recruiting | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC2435
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: proteomic; plasma proteomic; P16INK4A; chemotherapy; T cells; aging; morbidity
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected at two time points (pre-chemotherapy or shortly after breast cancer diagnosis if no chemotherapy is planned and then again 6-8 months later), plasma samples will be aliquoted and T cells will be separated and expression of p16INK4a mRNA in peripheral blood T-lymphocytes will be determined.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Chemotherapy: 40 patients with early-stage breast cancer whose treatment plan includes adjuvant or neoadjuvant chemotherapy.
  Interventions: Diagnostic Test: p16INK4a mRNA level assessment; Diagnostic Test: organ-specific protein signatures assessment
- Control: 20 patients with early-stage breast cancer whose treatment plan does not includeadjuvant or neoadjuvant chemotherapy.
  Interventions: Diagnostic Test: p16INK4a mRNA level assessment; Diagnostic Test: organ-specific protein signatures assessment

INTERVENTIONS:
Diagnostic Test: p16INK4a mRNA level assessment — Blood samples will be collected at two time points, plasma samples will be aliquoted, and T cells will be separated and expression of p16INK4a mRNA in peripheral blood T-lymphocytes will be determined
Diagnostic Test: organ-specific protein signatures assessment — Blood samples will be collected at two time points, plasma samples will be aliquoted, and organ-specific protein signatures assessment will be determined.

SUMMARY:
This study compares changes in P16INK4A expression and plasma proteomic signatures of specific organ age pre- and post-chemotherapy in women treated with adjuvant chemotherapy for early-stage breast cancer. It aims to determine if biological and accelerated immune aging, assessed using T cells from peripheral blood, represents aging in different organs.

Patients receiving chemotherapy, especially adjuvant regimens that include anthracyclines and taxanes, often experience late development of cardiac toxicity, functional loss, and cognitive decline. Comparing baseline characteristics with organ aging before therapy might identify patients at the highest risk for chemotherapy complications. For example, this is clinically significant for patients whose therapy includes taxanes or other drugs known to cause peripheral neuropathy. Identifying aging in the neurological or vascular systems before treatment might lead to changes in regimens.

Determining accelerated aging in specific organs allows for investigating interventions to mitigate organ damage. For instance, identifying patients at the highest risk of cardiac aging after treatment could lead to testing the effects of exercise, senolytics, and other strategies to reduce the risk of long-term heart disease.

DETAILED DESCRIPTION:
Chemotherapy has revolutionized cancer treatment, significantly improving relapse-free and survival rates for many cancers. However, these advances have come with a downside, and nowhere is this more evident than in childhood cancer. Despite the significant advances in the curability of most childhood cancers, up to 20% of patients die of comorbidity and secondary cancers by the age of 35 years.

Recent research shows that a plasma proteomic measure of protein abundance and expression can provide a" global" proteomic signature that accurately predicts chronologic age in the general population. It was shown that accelerated organ aging conferred a 20-50% higher mortality risk, and this was pronounced for those with accelerated cardiac and brain aging.

Previous studies have shown that p16INK4a, a robust biomarker of cell senescence measured in peripheral blood T cells, rises dramatically and likely irreversibly after adjuvant therapy for breast cancer. For anthracycline regimens, p16INK4a changes suggest 10 to 20 years of accelerated aging shortly after treatment. Additionally, in murine models, changes in P16INK4A are seen in all organs as mice age, but not all organs age at the same rate.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥22years and <66 years
* Diagnosed with early-stage breast cancer (The American Joint Committee on Cancer stages I-III).
* Understand and read English.
* Receive care at the study site.
* Able to understand and participate in study procedures for length of study.

Exclusion Criteria:

* Unable to provide consent, unable to communicate verbally.
* Unable to understand or read English.
* Enrolled in hospice care.

Ages: 22 Years to 66 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with breast carcinoma were treated at the study site. Groups will be stratified to ensure that those receiving anthracycline-containing regimens are well-represented and into three different age groups: < 50, 50 to 65, and 66 years and older
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
p16INK4a level changes over time | Up to 8 months
  The p16INK4a level will be determined from collected samples in each group. For the Chemotherapy Group, samples will be drawn before chemotherapy and 6-8 months after chemotherapy. For the Control Group, samples will be collected after diagnosis and again 6-8 months later. The differences will be tabulated.
Organ-specific protein expression change over time | Up to 8 months
  Organ-specific protein levels will be determined from collected samples in each group. For the Chemotherapy Group, samples will be drawn before chemotherapy and 6-8 months after chemotherapy. For the Control Group, samples will be collected after diagnosis and again 6-8 months later. The differences will be tabulated in grams per deciliter (g/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Hyman Muss, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials